CLINICAL TRIAL: NCT04408599
Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety and Tolerability Study of NC410 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: A Safety and Tolerability Study of NC410 in Subjects With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Upon completion of the Phase 1 portion of the NC410 monotherapy trial, NextCure focused efforts on a combination trial of NC410 in solid tumors.
Sponsor: NextCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NC410-01
Record Dates: First submitted 2020-05-19; First posted 2020-05-29 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Advanced or Metastatic Solid Tumors; Ovarian Cancer; Gastric Cancer; Colo-rectal Cancer
Keywords: Advanced Cancer; Metastatic Cancer; NC410; Solid Tumor; Immunotherapy; PK; Ovarian Cancer; Gastric Cancer; Colo-rectal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Stomach Neoplasms; Colonic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- NC410 3mg (Experimental): 3mg of NC410 for IV infusion administered in 14 day dosing cycles
  Interventions: Drug: NC410
- NC410 6mg (Experimental): 6mg of NC410 for IV infusion administered in 14 day dosing cycles
  Interventions: Drug: NC410
- NC410 15mg (Experimental): 15mg of NC410 for IV infusion administered in 14 day dosing cycles
  Interventions: Drug: NC410
- NC410 30mg (Experimental): 30mg of NC410 for IV infusion administered in 14 day dosing cycles
  Interventions: Drug: NC410
- NC410 60mg (Experimental): 60mg of NC410 for IV infusion administered in 14 day dosing cycles
  Interventions: Drug: NC410
- NC410 100mg (Experimental): 100mg of NC410 for IV infusion administered in 14 day dosing cycles
  Interventions: Drug: NC410
- NC410 200mg (Experimental): 200mg of NC410 for IV infusion administered in 14 day dosing cycles
  Interventions: Drug: NC410

INTERVENTIONS:
Drug: NC410 — NC410 is an experimental antibody drug that may make the immune response more active against cancer

SUMMARY:
This research study is studying a new drug, NC410, as a possible treatment for advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older.
* Willingness to provide written informed consent for the study.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Locally advanced or metastatic disease; locally advanced disease must not be amenable to resection with curative intent.
* Subjects who have disease progression after treatment with available therapies that are known to confer clinical benefit, or who are intolerant to treatment, or who refuse standard treatment. Note: There is no limit to the number of prior treatment regimens.
* Presence of measurable disease based on RECIST v1.1. Tumor lesions situated in a previously irradiated area, or in an area subjected to other locoregional therapy, are not considered measurable unless there has been demonstrated progression in the lesion.
* After dose escalation, subject must be willing to undergo pretreatment and on-treatment tumor biopsies (core or excisional). Note: A baseline biopsy obtained for other purposes (i.e., not an NC410-01 study procedure) before signing consent may be utilized if the subject has not had any intervening systemic therapy from the time of the biopsy to the start of treatment with the medical monitor's approval.
* Female subjects of childbearing potential (defined as women who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy and are not postmenopausal, defined as ≥ 12 months of amenorrhea) must have a negative serum pregnancy test at screening. All female and male subjects of childbearing potential must agree to take appropriate precautions to avoid pregnancy or fathering children (with at least 99% certainty) from screening through 60 days after the last dose of study drug.

Exclusion Criteria:

* Inability to comprehend or unwilling to sign the Informed Consent Form.
* Screening laboratory values of:

  1. Absolute neutrophil count < 1.5 × 10^9/L
  2. Platelets < 100 × 10^9/L
  3. Hemoglobin < 9 g/dL or < 5.6 mmol/L
  4. Serum creatinine > 1.5 × institutional upper limit of normal (ULN)
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 2.5 × ULN
  6. Total bilirubin ≥ 1.5 × ULN unless conjugated bilirubin ≤ ULN (conjugated bilirubin only needs to be tested if total bilirubin exceeds ULN). If there is no institutional ULN, then direct bilirubin must be < 40% of total bilirubin.
  7. International normalized ratio (INR) or prothrombin time (PT) > 1.5 × ULN
  8. Activated partial thromboplastin time (aPTT) > 1.5 × ULN
* Transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 14 days before the first administration of study drug.
* Receipt of anticancer medications or investigational drugs within the following intervals before the first administration of study drug:

  1. ≤ 14 days for chemotherapy, targeted small molecule therapy, or radiation therapy. Subjects must also not require chronic use of corticosteroids and must not have had radiation pneumonitis because of a treatment. A 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease with medical monitor approval. Note: Bisphosphonates and denosumab are permitted medications.
  2. ≤ 28 days for prior immunotherapy or persistence of active cellular therapy (e.g., chimeric antigen receptor T cell therapy; other cellular therapies must be discussed with the medical monitor to determine eligibility).
  3. ≤ 28 days for a prior monoclonal antibody used for anticancer therapy except for denosumab.
  4. ≤ 7 days for immune-suppressive-based treatment for any reason. Note: Use of inhaled or topical steroids or corticosteroid use for radiographic procedures is permitted. Note: The use of physiologic corticosteroid replacement therapy may be approved after consultation with the medical monitor.
  5. ≤ 28 days or 5 half-lives (whichever is longer) before the first dose for all other investigational study drugs or devices. For investigational agents with long half-lives (e.g., > 5 days), enrollment before the fifth half-life requires medical monitor approval.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy (including prior immunotherapy) and/or complications from prior surgical intervention before starting therapy. Note: Subjects with stable chronic conditions (≤ Grade 2) not expected to resolve (such as neuropathy and alopecia) are exceptions and may enroll. Note: Subjects with a history of any grade immune-related ocular AE (e.g., episcleritis, scleritis, uveitis) will be excluded.
* Receipt of a live vaccine within 30 days of planned start of study therapy. Note: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox/zoster, yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
* Active autoimmune disease that required systemic treatment in the past (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Subjects who have not required systemic treatment in the past 2 years may be eligible with approval of the medical monitor. Note: Subjects with hyper/ hypothyroidism are eligible to participate. Note: Replacement and symptomatic therapies (e.g., levothyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) are not considered a form of systemic immune suppressive therapy and are allowed.
* Known active CNS metastases and/or carcinomatous meningitis. Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 28 days before the first dose of study drug and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases or CNS edema, and have not required steroids for at least 7 days before the first dose of study drug.
* Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry apart from cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy, or cancers from which the subject has been disease-free for > 1 year, after treatment with curative intent.
* Evidence of active, noninfectious pneumonitis or history of interstitial lung disease.
* History or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful.
* Active infection requiring systemic therapy.
* Evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection or risk of reactivation. HBV-DNA and HCV-RNA must be undetectable. Subjects cannot be positive for HBV-DNA, HCV-RNA, hepatitis B surface antigen, or anti-hepatitis B core antibody. Note: Subjects with no prior history of hepatitis B infection who have been vaccinated against hepatitis B and who have a positive antibody against hepatitis B surface antigen test as the only evidence of prior exposure may participate in the study.
* Known history of HIV (HIV 1 or HIV 2 antibodies).
* Known allergy or reaction to any component of study drug or formulation components.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 60 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han Myint, MD, Study Director — NextCure, Inc.
Locations (5):
- United States (5):
  - NIH National Cancer Institute (NCI), Bethesda, Maryland
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Langone Health, New York, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UT MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 46 participants took part in the study at 5 investigative sites in the United States from 10Jun2020 to 06Jul2023.
Pre-assignment Details: Phase 1a (Dose Escalation) consisted of 7 planned cohorts (NC410 IV doses 3mg to 200mg). Phase 1b (Safety Expansion) consisted of 3 cohorts (NC410 IV doses 30mg , 60mg and 100mg). Phase 1 enrolled 46 participants. NextCure decided to forgoe moving forward with NC10 as a monotherapy in Phase 2.
Period: Overall Study
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
Started | 3 | 3 | 4 | 10 | 10 | 10 | 6
Completed | 1 | 2 | 1 | 7 | 7 | 6 | 1
Not Completed | 2 | 1 | 3 | 3 | 3 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg | Total
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 10 | 10 | 6 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (7.64) | 61.3 (13.32) | 59.0 (2.45) | 58.2 (14.44) | 66.3 (14.69) | 59.3 (9.46) | 66.0 (7.48) | 61.0 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 7 | 3 | 7 | 5 | 28
  Male | 1 | 1 | 2 | 3 | 7 | 3 | 1 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 3 | 3 | 2 | 10 | 10 | 9 | 5 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 3 | 4 | 2 | 1 | 11
  White | 2 | 3 | 4 | 5 | 5 | 7 | 4 | 30
  More than one race | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 4 | 10 | 10 | 10 | 6 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events as Assessed by CTCAE v5.0
Description: Number of Participants With Treatment-emergent Adverse Events
Time Frame: From enrollment through up to 90 days after end of treatment, an average of 1 year
Population: The Safety Analysis Set (SAS) will include all the subjects who receive any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 10 | 10 | 6
Participants | 3 | 3 | 4 | 9 | 10 | 9 | 6

2. Secondary Outcome: Objective Response Rate Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To assess antitumor activity/efficacy by evaluating objective response rate (ORR), defined as the percentage of participants who experienced a complete response (CR; disappearance of all target lesions) or a partial response (PR; at least a 30% decrease in the sum of diameters of target lesions) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC410.
Measure: Count of Participants; unit: Participants
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 10 | 10 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Duration of Response Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and Modified Response Evaluation Criteria in Solid Tumors
Description: To assess antitumor activity/efficacy by evaluating duration of response (DoR), defined as the time from the first documented complete response or partial response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Modified Response Evaluation Criteria in Solid Tumors to the first documented progressive disease or death due to any cause, whichever occurs first. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: CompleteResponse (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
  .
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC410.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 10 | 10 | 6
months | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.

4. Secondary Outcome: Disease Control Rate Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: To assess antitumor activity/efficacy by evaluating disease control rate (DCR), defined as the proportion of participants in whom a documented complete response, partial response, or stable disease is observed as the best overall response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: Approximately 1 year
Population: The FAS includes all subjects enrolled in the study who received at least one full dose of NC410
Measure: Count of Participants; unit: Participants
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 10 | 10 | 6
Participants | 1 | 3 | 1 | 1 | 1 | 1 | 1

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of NC410
Description: To evaluate the Maximum Plasma Concentration (Cmax) of NC410
Time Frame: Days 1, 2, 3 and 8 of Cycles 1 and 5. Each cycle is 14 days in duration.
Population: The PK analysis set (PAS) will include all the subjects whose blood samples are collected for PK analysis.
  One subject within NC410 100mg Arm/Group has been excluded from the summary table due to the day 1 pre-infusion and post-infusion concentration values being incorrect
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
Number analyzed (Participants) | 0 | 0 | 4 | 10 | 10 | 9 | 6
ng/mL
  Cycle 1 |  |  | NA (NA) — The mean and SD were below lower limit of detection | 754 (295) | 2801 (1102) | 5296 (4405) | 11665 (9821)
  Cycle 5: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 1 | 1
  Cycle 5 |  |  | 443 (NA) — SD was below lower limit of detection | 1490 (184) | 2200 (NA) — SD was below lower limit of detection | 2220 (NA) — SD was below lower limit of detection | 2880 (NA) — SD was below lower limit of detection

6. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and Modified Response Evaluation Criteria in Solid Tumors
Description: To evaluate progression-free survival (PFS), defined as the time from the first dose of NC410 to the first occurrence of documented progressive disease or death due to any cause, whichever occurs first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), asa 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
  .
Time Frame: Approximately 1 year
Population: The FAS includes all subjects enrolled in the study who received at least one full dose of NC410
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 10 | 10 | 6
Months | 1.7 [1.6 to NA] — The upper limit of the confidence interval were not estimable due to limited number of participants with events. | 3.6 [3.6 to NA] — TThe upper limit of the confidence interval were not estimable due to limited number of participants with events. | 1.3 [0.5 to NA] — The upper limit of the confidence interval were not estimable due to limited number of participants with events. | 1.7 [1.0 to 3.5] | 1.4 [1.0 to 1.7] | 1.4 [1.2 to 1.8] | 1.8 [1.2 to NA] — The upper limit of the confidence interval were not estimable due to limited number of participants with events.

7. Secondary Outcome: Overall Survival (OS) as Assessed by Time of Death
Description: To evaluate overall survival (OS), defined as the time from the first dose of NC410 to death due to any cause.
Time Frame: Approximately 1 year
Population: The full analysis set (FAS) includes all subjects enrolled in the study who received at least one full dose of NC410.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
Number analyzed (Participants) | 3 | 3 | 4 | 10 | 10 | 10 | 6
months | NA [7.6 to NA] — The median and upper limit of the confidence interval were not estimable due to limited number of participants with event. | 5.3 [4.1 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with event. | NA [NA to NA] — The median and confidence intervals were not estimable due to limited number of participants with event. | NA [1.4 to NA] — The median and upper limit of the confidence interval were not estimable due to limited number of participants with event. | 4.8 [1.0 to NA] — The upper limit of the confidence interval was not estimable due to limited number of participants with event. | NA [1.3 to NA] — The median and upper limit of the confidence interval were not estimable due to limited number of participants with event. | NA [1.2 to NA] — The median and upper limit of the confidence interval were not estimable due to limited number of participants with event.

8. Secondary Outcome: Area Under the Curve (AUC) of NC410
Description: To evaluate the Area Under the Curve (AUC) of NC410.
Time Frame: Days 1, 2, 3 and 8 of Cycles 1 and 5. Each cycle is 14 days in duration.
Population: The PK analysis set (PAS) will include all the subjects whose blood samples are collected for PK analysis. AUC to Last Nonzero concentration.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
Number analyzed (Participants) | 0 | 0 | 4 | 10 | 10 | 10 | 6
h*ng/mL
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 10 | 10 | 9 | 6
  Cycle 1 |  |  |  | 13528 (15259) | 64530 (38613) | 107591 (52432) | 263894 (121831)
  Cycle 5: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 1 | 1
  Cycle 5 |  |  | 1056 (NA) — Standard Deviation was below the lower limit of detection | 47324 (3674) | 41448 (NA) — Standard Deviation was below the lower limit of detection | 205493 (NA) — Standard Deviation was below the lower limit of detection | 260199 (NA) — Standard Deviation was below the lower limit of detection

9. Secondary Outcome: Half-life (t1/2) of NC410
Description: To evaluate the half-life (t1/2) of NC410
Time Frame: Days 1, 2, 3 and 8 of Cycles 1 and 5. Each cycle is 14 days in duration.
Population: The PK analysis set (PAS) will include all the subjects whose blood samples are collected for PK analysis. Half-Life Lambda z (h).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
Number analyzed (Participants) | 0 | 0 | 4 | 10 | 10 | 10 | 6
hours
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 8 | 10 | 5 | 6
  Cycle 1 |  |  |  | 75.7 (74.7) | 126 (52.0) | 173 (43.6) | 111 (53.8)
  Cycle 5: number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 1 | 1
  Cycle 5 |  |  |  | 138 (7.23) | 41.1 (NA) — Standard Deviation was below the lower limit of detection | 156 (NA) — Standard Deviation was below the lower limit of detection | 194 (NA) — Standard Deviation was below the lower limit of detection

ADVERSE EVENTS:
Time Frame: From enrollment through up to 90 days after end of treatment, an average of 1 year.
Description: The severity of AEs will be assessed using NCI CTCAE v5.0 Grades 1 through 4. The NCI CTCAE v5.0 severity of Grade 5 will not be used; AEs resulting in death will be graded accordingly using Grades 1 through 4 and have theoutcome noted as fatal.
Arm/Group | NC410 3mg | NC410 6mg | NC410 15mg | NC410 30mg | NC410 60mg | NC410 100mg | NC410 200mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/3 | 0/4 | 2/10 | 4/10 | 3/10 | 1/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 2/4 | 5/10 | 5/10 | 7/10 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 9/10 | 10/10 | 9/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NC410 3mg (N=3) | NC410 6mg (N=3) | NC410 15mg (N=4) | NC410 30mg (N=10) | NC410 60mg (N=10) | NC410 100mg (N=10) | NC410 200mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Disease Progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic Haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion Related Hypersensitivity reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral Ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NC410 3mg (N=3) | NC410 6mg (N=3) | NC410 15mg (N=4) | NC410 30mg (N=10) | NC410 60mg (N=10) | NC410 100mg (N=10) | NC410 200mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 3 | 6 | 5 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 3 | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 4 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 4 | 4 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 3 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 2 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related hypersensitivity reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 3 | 2 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stoma prolapse (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1 | 1 | 1 | 2 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 3 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 3 | 0 | 2 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 2 | 0 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 2 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 4 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 4 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish study results before the first multi-center publication. If a multi-center publication is not submitted within 12 months after the end of the study at all sites, or if Sponsor confirms there will be no multi-center publication, the PI may publish study results. However, PI will allow Sponsor at least 30 days to review any publication of study results and Sponsor may request an additional 60 days to review the publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT04408599/Prot_SAP_000.pdf